CLINICAL TRIAL: NCT01522287
Title: Computer Assisted CBT for OCD: A Comprehensive Stepped-Care Approach
Brief Title: Computer Assisted Cognitive Behavior Therapy for Obsessive Compulsive Disorder: A Comprehensive Stepped-Care Approach
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Center for Psychological Consultation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R43MH090612 (NIH)
Record Dates: First submitted 2012-01-23; First posted 2012-01-31 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Obsessive Compulsive Disorder; Computer Assisted Therapy; Cognitive Behavior Therapy; Cognitive Therapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Behavior Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BT STEPS alone (Active Comparator): Subjects assigned to BT STEPS without coaching will receive computer assisted Cognitive Behavior Therapy. They will receive a welcome and orientation call from the project manager and up to three automated reminder e-mails if there is no activity in the BT Steps website for 5 days. E-mails will describe most recent "step" the participant used and what to expect in upcoming steps. The focus of reminder messages is on the patient"s progress through BT STEPS.
  Interventions: Behavioral: Computer-Assisted Cognitive Behavior Therapy (BT STEPS)
- BT Steps with non-therapist coaching (Active Comparator): Subjects randomized to BT STEPS with coaching will receive computer assisted Cognitive Behavior Therapy plus regularly scheduled weekly coaching, encouragement and support via phone. Calls will focus on user's progress in BT STEPS, troubleshoot problems the participant is having with the program, and set progress goals for the next coaching session. Coaches will be supervised by the CBT therapist, and may consult with the CBT clinician as needed.
  Interventions: Behavioral: Computer-Assisted Cognitive Behavior Therapy (BT STEPS)
- BT STEPS with therapist coaching (Active Comparator): Subjects randomized to BT STEPS with therapist coaching will receive computer-assisted Cognitive Behavior Therapy plus regularly scheduled weekly coaching and support from a CBT therapist via phone. Calls will focus on user's progress in BT STEPS, troubleshoot problems the participant is having with the program, and set progress goals for the next coaching session.
  Interventions: Behavioral: Computer-Assisted Cognitive Behavior Therapy (BT STEPS)

INTERVENTIONS:
Behavioral: Computer-Assisted Cognitive Behavior Therapy (BT STEPS) — BT STEPS is a computer-assisted self help treatment for OCD. Clients work through the program at their own pace.
  Other Names: Cogntive Therapy; Behavior Therapy; Cognitive-Behavior Therapy

SUMMARY:
The goal of this project is to improve access to effective treatments for obsessive compulsive disorder (OCD) through the use of web-based cognitive behavioral therapy (CBT) treatment. There intervention involves both a computer program (BT Steps) and human interaction via telephone. The investigators will test the efficacy and feasibility of computer therapy alone (n=35), computer plus a non-therapist coach (n=35), and computer plus a CBT therapist coach (n=35

DETAILED DESCRIPTION:
The need for evidence-based mental health treatments i.e., 'treatment based on the best available science or research evidence"1, has been stressed from scientific, ethical, and marketing perspectives. While empirical evidence supports both the efficacy and effectiveness of cognitive behavior therapy (CBT) for Obsessive-Compulsive Disorder (OCD), demand for clinicians trained in these approaches far exceeds supply. New technologies provide the opportunity to facilitate access to this specialized treatment. A growing body of research has found that web-based self-administered psychotherapy is highly effective, cost-efficient, and can achieve clinical improvements similar to those obtained with clinician administered therapy. The long-term goal of this project is to improve clinical and occupational functioning and decrease disability associated with OCD by improving access to effective treatments through the use of web-based CBT treatment. The intervention involves a computer program (BT STEPS) and human interaction via telephone. The inclusion of human interaction for coaching and encouragement has been found to significantly increase compliance and success rates in computerized self-help. Whether treatment outcomes differ when this coaching is done by a therapist versus when done by a trained non-therapist has not been studied. This is the first program to examine a hybrid model involving different levels of remote clinician coaching in combination with an on-line self-help tutorial. In Phase I the investigators will test the efficacy and feasibility of computer therapy alone (n=35), computer plus nontherapist coach (n=35) and computer plus CBT therapist coach. In phase II the investigators will do a fully powered study comparing our model to traditional face-to-face therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* Have clinically significant OCD
* YBOCS score of 16-32

Exclusion Criteria:

* Significant comorbid depression
* Serious suicide risk
* Psychosis or psychotic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale (YBOCS) | Change from Baseline on YBOCS at 12 weeks
  YBOCS measures severity of obsessions and compulsions

SECONDARY OUTCOMES:
PHQ-9 | Change from baseline on PHQ9 at 12 weeks
  PHQ-9 assesses the 9 core DSM symptoms of depression
Work and Social Adjustment Scale (WSA) | Change from baseline on WSA at 12 weeks
  Measures problems at work and social relationships

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Psychological Consultation, Madison, Wisconsin, United States

REFERENCES:
- [Background] Greist JH, Marks IM, Baer L, Kobak KA, Wenzel KW, Hirsch MJ, Mantle JM, Clary CM. Behavior therapy for obsessive-compulsive disorder guided by a computer or by a clinician compared with relaxation as a control. J Clin Psychiatry. 2002 Feb;63(2):138-45. doi: 10.4088/jcp.v63n0209. PMID 11874215